CLINICAL TRIAL: NCT03390218
Title: Comparison of Treatment for Anxiety and Depression Augmented With TAO to Treatment as Usual (TAU) in the Weber Human Services
Brief Title: TAO Outpatient Trial for Anxiety and Depression
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: TAO Connect, Inc. (Industry)
Responsible Party: Principal Investigator, Sherry Benton, Chief Science Officer, TAO Connect, Inc.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TAO001
Record Dates: First submitted 2017-11-27; First posted 2018-01-04 (Actual); Last update posted 2018-01-04 (Actual); Status verified 2018-01

CONDITIONS: Anxiety Disorders; Depression
MeSH Terms: conditions — Anxiety Disorders; Depression | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: Randomized control trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TAO (Therapy Assisted Online) (Experimental): TAO participants will attend a once weekly group in a computer lab. Each participant will complete an interactive educational module using an evidence based protocoled treatment for anxiety and/or depression, and have a brief session with the group leader to discuss application of the content. Participants will have access to a companion app they may use between sessions to practice skills and reinforce learning.
  Interventions: Behavioral: Therapy Assistance Online
- Treatment as usual (Active Comparator): After the completion of a psychosocial assessment, and development of a treatment plan, clients are offered individual and group therapy sessions, case management services, and medication management services depending on the diagnoses. Individual and group therapy is often generic in nature as well, although some structured, evidence-based treatments are offered such as Psycho-Education Multi-Family Group and Illness Management Recovery.
  Interventions: Behavioral: Treatment as usual

INTERVENTIONS:
Behavioral: Therapy Assistance Online — protocoled on-line educational modules, with brief therapist interaction and practice support with a mobile app.
  Arms: TAO (Therapy Assisted Online)
Behavioral: Treatment as usual — Individual and group therapy, generic in nature
  Arms: Treatment as usual

SUMMARY:
Access to effective treatment resources is a ubiquitous problem in behavioral health. There is a need for effective interventions that are more easily accessed at a lower cost. This study will compare outcomes for two models of treatment: 1) The experimental group, Therapy Assistance Online (TAO), and 2) the comparison group, treatment as usual.

DETAILED DESCRIPTION:
Access to effective treatment resources is a ubiquitous problem in behavioral health. There is a need for effective interventions that are more easily accessed at a lower cost. This stud will compare outcomes for two models of treatment: 1) The experimental group, Therapy Assistance Online (TAO), and 2) the comparison group, treatment as usual.

TAO group TAO is a suite of tools for providing patient education, support, and accountability delivered digitally. Educational materials are organized in an evidence based-protocolled treatment for anxiety or depression. TAO participants will attend a once weekly group in a computer lab. Each participant will complete an interactive educational module and have a brief session with the group leader to discuss application of the content. Participants will have access to a companion app they may use between sessions to practice skills and reinforce learning.

Treatment as Usual Group - After the completion of a psychosocial assessment, and development of a treatment plan, clients are offered individual and group therapy sessions, case management services, and medication management services depending on the diagnoses. Individual and group therapy is often generic in nature as well, although some structured, evidence-based treatments are offered such as Psycho-Education Multi-Family Group and Illness Management Recovery.

Potential participants will receive an initial evaluation and screening to determine diagnosis, appropriateness for the study, and level of care required. Informed consent will include a statement indicating that agreement to participate will not affect access to treatment. Those who do not wish to participate will receive care as usual. Patients who agree to participate will be randomly assigned to either treatment as usual or treatment augmented with TAO.

Referral and Randomization Process -

1. Therapist identifies a client who meets the inclusionary criteria.
2. Clinician explains the availability of the TAO support services and the current study and invites the client to participate.
3. If the client agrees to participate, the clinician will explain the study and have the client sign the consent to participate form and call customer care to determine if the client will be in the experimental group (A) or control group (B).
4. If client is assigned to the experimental group, the clinician will help the client select a time to participate in the TAO support services each week. The clinician will again explain the benefits of participation, seek a commitment to attend, and help resolve any ambivalence of the client to participate.
5. If client is assigned to treatment as usual, the clinician will help the client select a time to participate in group session.
6. The referring clinician will then email the group therapist to inform him/her of the referral.

Introducing the TAO Support Services to Potential Clients -

1. Ask permission to share information about the TAO Support Services
2. Explain that the TAO system provides mental health services through an electronic system completed on a computer. Clients watch videos and complete modules on a computer for approximately 45 minutes to an hour, one time each week for 8 weeks.
3. Explain that participation in these support services has been shown in other studies to reduce symptoms, and that a current study is underway to determine if this will prove helpful to clients at WHS.
4. Invite the client to participate in the study letting him/her know that agreeing to participate in the study does not guarantee access to the TAO system.
5. If client agrees -

   1. Have client sign the consent to participate form.
   2. Contact customer care to find out if the client is assigned to the TAO system or the control group.
6. If assigned to the TAO system, help the client know when and where to meet for the TAO session. Contact the group leader with client information.

Measures

Participants in both the experimental group (TAO) and the control group treatment as usual (TAU) will complete the OQ-45 at intake, and in each subsequent session. TAO participants will also complete the Behavioral Health Measure-20 just prior to each group session on the computer in the computer lab.

Participants in both the experimental group (TAO) and the control group (TAU) will complete the OQ-45 at intake and at each group session. WE Well-being scale.

Sessions completed. Demographics.

Subjects

Subjects will be clients seeking treatment for anxiety and depression at Weber Human Services. All participants will be adults (18 and over) who meet inclusion criteria. Clients who agree to participant will be randomly assigned to a treatment condition. We will enroll fifty clients per treatment condition and enrollment will be ongoing until the number is reached. Active treatment will be 8 weeks, with follow-up at 3 months. Participants will not receive renumeration for participation.

Researchers at (TAO Connect, Inc.) TCI will have no direct contact with the subjects. All data collection will occur through the computer system. TCI technical support staff will have minimal PHI: name, login, email address if the client requires any technical support.

ELIGIBILITY:
Inclusion Criteria:

* Clients in their first month of treatment with any primary or secondary diagnosis of depression or anxiety. This includes all forms of depression and/or anxiety disorder.

Exclusion Criteria:

* Chronic depression with a Likely Utilization of Services Instrument (LUSI) designation of "high" or "consistent user" of services. These clients should be referred to Illness Management Recovery.
* Clients with schizophrenia, or any other form of active psychosis.
* Clients with substance dependence disorder.
* Clients with personality disorders.
* Clients whose intellectual functioning would prevent understanding the TAO system and materials.
* Client must not have been in treatment for anxiety and depression in the past three months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2018-01-15 (Estimated); Primary Completion 2018-11 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Outcome Questionnaire-45 | At intake, 8 weeks, 12 weeks- change in scores
  45 question survey, assessing symptom change, the OQ-45 is the most commonly used measure of change in psychotherapy. The OQ-45 has one general scale and 3 sub-scales.
  1. The symptom distress scale scores range from 0-100 with a clinical cut-off of 36. Reliable change is indicated when a client's score changes by 10 points or more.
  2. The Interpersonal relations scale scores range from 0-44, the clinical cut-off is 15, reliable change when a client's score changes by 8 points or more.
  3. Social role scale, scores range from 0-36, clinical cut-off is 12 or more, reliable change is a change of 7 points or more

CONTACTS AND LOCATIONS:
Locations (1):
- Weber Human Services, Ogden, Utah, United States

IPD SHARING:
Plan to Share IPD: No
Sharing individual participant data in behavioral health is prohibited by law.